CLINICAL TRIAL: NCT03871569
Title: Medico-economical Evaluation on Buccodental Teleexpertise in Nursing Home
Acronym: e-DENT-EHPAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting and follow-up due to the epidemic context of COVID19
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL18_0079
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Tooth Diseases
Keywords: Telemedicine; dentistry; long-term-care-home
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telemedecine nursing home (Active Comparator): One buccodental teleexpertise at the completion day and a second buccodental teleexpertise at the end of study
  Interventions: Other: bucco-dental teleexpertise
- control nursing home (No Intervention): Only one buccodental teleexpertise at the end of study

INTERVENTIONS:
Other: bucco-dental teleexpertise — A bucco-dental consultation remotely using telemedicine system
  Arms: telemedecine nursing home

SUMMARY:
Oral care in medical and social institutions is a real public health problem. The impact of poor oral health on the general state of residents but also on their overall quality of life is significant.

The development of a precise regulatory framework for telemedicine in France aims to transform experiments into sustainable medical activities. Odontology often set aside in this reflection, must be reintegrated. The use of tele-expertise for the oral care of nursing home residents should make it possible to replace oral health in medico-social institutions. The investigators will assess in a cluster randomized controlled study whether the buccodental telemedicine has a viable economic model and a significant impact on the overall health of facility for dependent elderly persons residents.

The medico-economic impact of the buccodental telexpertise is fundamental for the development of this innovative activity.

ELIGIBILITY:
Inclusion Criteria:

* Be resident of a facility for dependent elderly persons involved in the study
* Have given their Free, informed and signed consent
* Beneficiary or member of a social security scheme

Exclusion Criteria:

* incapacity to open the mouth
* contrary opinion of the medical team (end of life)
* Change of nursing home planned within 6 months
* Subject in a period of relative exclusion from another protocol
* Subject's participation in another study
* Subject deprived of liberty by judicial or administrative decision

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Cost-Utility ratio of buccodental telemedicine in nursing home as compared to usual care | At month 6
  Costs include telemedicine and medical costs related to oral health care. Utility correspond to the Quality Adjusted Life-Years (QALY) score measured using the EQ5D-3L questionnaire (EuroQol 3 levels of 5 dimensions).

SECONDARY OUTCOMES:
Cost/Efficacity ratio of buccodental telemedicine in nursing home as compared to usual care | At month 6
  Costs include telemedicine and medical costs related to oral health care.
  The clinical efficacy criteria correspond to the proportion of patients with a zero dental emergency score. The score of Emergency is measured according to WHO classification:
  Score "0" correspond to "unnecessary care"
  Score "1" correspond to "descaling required"
  Score "2" correspond to "Low urgency: need for restoration and/or crown but not immediately (superficial damage to the tooth). Includes patients requiring fixed and/or removable prostheses".
  Score "3" correspond to: "Advanced emergency: need for restorations and/or crowns quickly (within 7 to 14 days) to avoid pulp damage and/or infection"
  Score "4" correspond to: "High urgency: urgent need for care due to pain and/or infection. Includes patients requiring endodontic treatment or extraction"
Quality of life comparison: EQ5D-3L questionnaire | At month 6
  The Quality of Life measured using the EQ5D-3L (EuroQol 3 levels of 5 dimensions) questionnaire. EQ-5D-3L questionnaire comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. Levels of perceived problems are coded as follows: Level 1 (no problems) is coded as a '1' - Level 2 (some problems) is coded as a '2' - Level 3 (extreme problems) is coded as a '3'. The best score for the 5 dimensions is coded by '11111' and the worst state is coded by '33333'. In addition a EQ visual analogue scale (EQ VAS) help people say how good or bad a health state is, on which the best state is marked 100 and the worst state is marked 0.
Economic impact of teleexpertise on dental treatment | At month 6
  Budgetary impact of the new coverage expressed in annual cash flows
Evaluate satisfaction rate of use of teleexpertise of nursing home staff | At month 6
  Satisfaction of nursing home staff measured by an ad hoc Likert scale
Compare the emergency score | At month 0 and at month 6
  The emergency score measured by the Oral Health Assessment Tool (OHAT) questionnaire. The OHAT comprises eight categories of screening tool to assess oral health : Lips, Tongue, Gums and tissues, Saliva, Natural teeth, Dentures, Oral cleanliness, Dental pain. After a dental examination by telemedicine, the dentist will evaluate each category as following : Score "0" correspond to "healthy", score "1" corresponds to "changes" or score "3" correspond to "unhealthy".

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Giraudeau, DDS, MSc, Principal Investigator — CHU de Montpellier
Locations (13):
- France (13):
  - EHPAD Le Sherpa, Belmont-sur-Rance
  - EHPAD Via Domitia, Castelnau-le-Lez
  - EHPAD Korian La Colombe, Gigean
  - EHPAD Korian Perier, Marseille
  - EHPAD La Roselière, Marsillargues
  - EHPAD Françoise Gauffier, Montpellier
  - EHPAD Korian La Pompignane, Montpellier
  - EHPAD La Carriera, Montpellier
  - EHPAD Montpellieret, Montpellier
  - EHPAD Pierre Laroque, Montpellier
  - Résidence mutualiste de Pezilla, Pezilla La Rivière
  - EHPAD Saint Jean, Saint-Amans-des-Cots
  - EHPAD Saint Jean Pla de Corts, St. Jean-Pla-de-Corts

IPD SHARING:
Plan to Share IPD: No